CLINICAL TRIAL: NCT02516046
Title: A Clinico-Pathological Study of the Correspondence Between 18F-AV-1451 PET Imaging and Post-Mortem Assessment of Tau Pathology
Brief Title: 18F-AV-1451 Autopsy Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A16
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2020-09-07 (Actual); Last update posted 2020-09-07 (Actual); Status verified 2020-09

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Flortaucipir PET Scan (Experimental)
  Interventions: Drug: Flortaucipir F18; Procedure: PET Scan

INTERVENTIONS:
Drug: Flortaucipir F18 — 370 megabecquerel (MBq) IV single-dose
  Other Names: [F-18]T807; 18F-AV-1451; LY3191748
Procedure: PET Scan — positron emission tomography (PET) scan

SUMMARY:
This study is designed to test the relationship between ante-mortem flortaucipir Positron Emission Tomography (PET) imaging and tau neurofibrillary pathology associated with Alzheimer's disease (AD), as measured at autopsy.

ELIGIBILITY:
Inclusion Criteria:

* Have a projected life expectancy of ≤ 6 months
* Can tolerate a 20 minute PET scan
* Give informed consent or have a legally authorized representative to consent for study procedures and brain donation consistent with the legal requirements of the State in which they die

Exclusion Criteria:

* Aggressively being treated with life sustaining measures
* Known to have a structural brain lesion that would interfere either with PET imaging or pathological assessment
* Clinically significant infectious disease
* Currently receiving any investigational medications except with permission from the study sponsor
* Participated in an experimental study with an amyloid or tau targeting agent
* Suspected encephalopathy due to alcoholism or end-stage liver disease
* Females of childbearing potential
* History of risk factors for Torsades de Pointes or are currently taking medication known to cause QT prolongation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-09; Primary Completion 2018-06-13 (Actual); Study Completion 2018-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Chair — Avid Radiopharmaceuticals, Inc.
Locations (31):
- United States (30):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Cherlin Research, Los Gatos, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - California Research Foundation, San Diego, California
  - Pacific Research Network, San Diego, California
  - Ray Dolby Brain Health Center, San Francisco, California
  - Syrentis Clinical Research, Santa Ana, California
  - Neuropsychiatric Research Center of Southwest Florida, Fort Myers, Florida
  - Galiz Research, Hialeah, Florida
  - Merritt Island Medical Research, Merritt Island, Florida
  - Miami Jewish Health Systems, Miami, Florida
  - D de la Vega MD Research Group, Miami, Florida
  - Bioclinica, Orlando, Florida
  - Emory University Brain Health Center, Atlanta, Georgia
  - Alzheimer's Disease Center, Quincy, Massachusetts
  - Steinberg Diagnostics, Henderson, Nevada
  - Adirondack Medical Research Center, Glens Falls, New York
  - Clarity Clinical Research, LLC, Syracuse, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Valley Medical Primary Care, Centerville, Ohio
  - Hospice of the Western Reserve, Cleveland, Ohio
  - American Clinical Trials, LLC (Site 1216), Oklahoma City, Oklahoma
  - Oklahoma Behavioral Health, Oklahoma City, Oklahoma
  - Rhode Island Hospital, Providence, Rhode Island
  - Houston Methodist Research Institute, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - Overlake Internal Medicine Associates, PS, Bellevue, Washington
  - University of Washington Medicine, Seattle, Washington
- University of Melbourne, Parkville, Victoria, Australia

REFERENCES:
- [Background] Hyman BT, Phelps CH, Beach TG, Bigio EH, Cairns NJ, Carrillo MC, Dickson DW, Duyckaerts C, Frosch MP, Masliah E, Mirra SS, Nelson PT, Schneider JA, Thal DR, Thies B, Trojanowski JQ, Vinters HV, Montine TJ. National Institute on Aging-Alzheimer's Association guidelines for the neuropathologic assessment of Alzheimer's disease. Alzheimers Dement. 2012 Jan;8(1):1-13. doi: 10.1016/j.jalz.2011.10.007. PMID 22265587
- [Background] Montine TJ, Phelps CH, Beach TG, Bigio EH, Cairns NJ, Dickson DW, Duyckaerts C, Frosch MP, Masliah E, Mirra SS, Nelson PT, Schneider JA, Thal DR, Trojanowski JQ, Vinters HV, Hyman BT; National Institute on Aging; Alzheimer's Association. National Institute on Aging-Alzheimer's Association guidelines for the neuropathologic assessment of Alzheimer's disease: a practical approach. Acta Neuropathol. 2012 Jan;123(1):1-11. doi: 10.1007/s00401-011-0910-3. Epub 2011 Nov 20. PMID 22101365
- [Result] Fleisher AS, Pontecorvo MJ, Devous MD Sr, Lu M, Arora AK, Truocchio SP, Aldea P, Flitter M, Locascio T, Devine M, Siderowf A, Beach TG, Montine TJ, Serrano GE, Curtis C, Perrin A, Salloway S, Daniel M, Wellman C, Joshi AD, Irwin DJ, Lowe VJ, Seeley WW, Ikonomovic MD, Masdeu JC, Kennedy I, Harris T, Navitsky M, Southekal S, Mintun MA; A16 Study Investigators. Positron Emission Tomography Imaging With [18F]flortaucipir and Postmortem Assessment of Alzheimer Disease Neuropathologic Changes. JAMA Neurol. 2020 Jul 1;77(7):829-839. doi: 10.1001/jamaneurol.2020.0528. PMID 32338734
- [Derived] Pontecorvo MJ, Keene CD, Beach TG, Montine TJ, Arora AK, Devous MD Sr, Navitsky M, Kennedy I, Joshi AD, Lu M, Serrano GE, Sue LI, Intorcia AJ, Rose SE, Wilson A, Hellstern L, Coleman N, Flitter M, Aldea P, Fleisher AS, Mintun MA, Siderowf A. Comparison of regional flortaucipir PET with quantitative tau immunohistochemistry in three subjects with Alzheimer's disease pathology: a clinicopathological study. EJNMMI Res. 2020 Jun 15;10(1):65. doi: 10.1186/s13550-020-00653-x. PMID 32542468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment occurred between October 2015 and June 2018. Enrolled end-of-life subjects (life expectancy less than 6 months) at hospice centers in the US and Australia consented to a flortaucipir PET scan and to brain donation at autopsy.
Pre-assignment Details: To be considered eligible for the primary analysis, death had to occur within 9 months of flortaucipir scan and valid autopsy was required. The first 3 subjects to come to autopsy were considered front-runners. Front-runner scan and autopsy results were unblinded to the sponsor to optimize analysis.
Groups:
- All Enrolled Cohort: End-of-life subjects consenting to brain donation at autopsy from the flortaucipir PET scan arm
Period: Overall Study
Arm/Group | All Enrolled Cohort
Started | 156 (Total number of subjects scanned)
Died While on Study | 73
Valid Autopsy Results and PET Scan | 67 (includes 3 front-runners)
Completed | 64 (Completed = included in autopsy cohort)
Not Completed | 92

BASELINE CHARACTERISTICS:
Groups:
- All Enrolled Cohort: All subjects consenting to flortaucipir PET and brain donation at autopsy
Arm/Group | All Enrolled Cohort
Number analyzed (Participants) | 156
Age, Continuous [Mean (Standard Deviation); unit: years] | 80.2 (12.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 86
  Male | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 136
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 143
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 151
  Australia | 5

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome 1: Diagnostic Performance of Individual Readers (NFT Score)
Description: Sensitivity and specificity of 5 independent readers' interpretations of ante-mortem flortaucipir PET imaging for detection of a pattern of flortaucipir neocortical uptake that corresponds to neurofibrillary tangles (NFT) Score of B3 (Hyman et al., 2012; Montine et al., 2012). NFT B scores range from B0 (Braak Stage 0; no NFTs in the brain) to B3 (Braak Stage V/VI; widespread NFTs in the brain). Sensitivity and specificity are percentages that can range from 0 to 100%. The hypothesis tested was that, of the 5 independent imaging physicians, at least 3 will have the lower bounds of 2-sided 95% CIs ≥50%, for both sensitivity and specificity.
Time Frame: at autopsy within 9 months of baseline scan
Population: Autopsy cohort N=64. n=39 were truth positive for NFTs. n=25 were truth negative for NFTs.
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Sensitivity of Flortaucipir vs Autopsy NFT Score B3: Subjects with a positive autopsy NFT score truth standard (NFT B3)
- Specificity of Flortaucipir vs Autopsy NFT Score <B3: Subjects with a negative autopsy NFT score truth standard (NFT B2 or lower)
Arm/Group | Sensitivity of Flortaucipir vs Autopsy NFT Score B3 | Specificity of Flortaucipir vs Autopsy NFT Score <B3
Number analyzed (Participants) | 39 | 25
percentage of cases correctly identified
  Reader 1 | 97.4 [86.8 to 99.5] | 68.0 [48.4 to 82.8]
  Reader 2 | 92.3 [79.7 to 97.3] | 92.0 [75.0 to 97.8]
  Reader 3 | 92.3 [79.7 to 97.3] | 88.0 [70.0 to 95.8]
  Reader 4 | 92.3 [79.7 to 97.3] | 76.0 [56.6 to 88.5]
  Reader 5 | 100 [91.0 to 100.0] | 52.0 [33.5 to 70.0]

2. Primary Outcome: Primary Outcome 2: Diagnostic Performance of Individual Readers (NIA-AA Autopsy Diagnosis)
Description: Sensitivity and specificity of 5 independent readers' interpretations of ante-mortem flortaucipir imaging for detection of a pattern of flortaucipir neocortical uptake that corresponds to high levels of Alzheimer's disease neuropathologic change (High ADNC) as defined by National Institute on Aging-Alzheimer's Association (NIA-AA) criteria. ADNC categories are None, Low, Intermediate and High, with High indicating the most severe level of AD-related pathology changes in the brain (Hyman et al., Alzheimers Dement. 2012 Jan;8(1):1-13). The hypothesis tested was that, of the 5 independent imaging physicians, at least 3 will have the lower bounds of 2-sided 95% CIs ≥50%, for both sensitivity and specificity.
Time Frame: at autopsy within 9 months of baseline scan
Population: Autopsy cohort N=64. n=38 were truth positive for NFTs. n=26 were truth negative for NFTs.
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Sensitivity of Flortaucipir vs NIA-AA Autopsy Diagnosis: Subjects with a positive truth standard (High ADNC)
- Specificity of Flortaucipir vs NIA-AA Autopsy Diagnosis: Subjects with a negative truth standard (No/Low/Intermediate ADNC)
Arm/Group | Sensitivity of Flortaucipir vs NIA-AA Autopsy Diagnosis | Specificity of Flortaucipir vs NIA-AA Autopsy Diagnosis
Number analyzed (Participants) | 38 | 26
percentage of cases correctly identified
  Reader 1 | 97.5 [87.1 to 99.6] | 65.4 [46.2 to 80.6]
  Reader 2 | 95.0 [83.5 to 98.6] | 92.3 [75.9 to 97.9]
  Reader 3 | 95.0 [83.5 to 98.6] | 88.5 [71.0 to 96.0]
  Reader 4 | 95.0 [83.5 to 98.6] | 76.9 [57.9 to 89.0]
  Reader 5 | 100 [91.2 to 100.0] | 50.0 [32.1 to 67.9]

3. Secondary Outcome: Flortaucipir Diagnostic Performance (NFT Score)
Description: Sensitivity and specificity of majority interpretation of AD pattern tau PET scan corresponding to NFT Score of B3. The 95% confidence intervals (CI) provided for specificity and sensitivity were based on the Wilson score method. The hypothesis tested was that majority read results had the lower bound of the 2-sided 95% CI greater than or equal to 55% for both sensitivity and specificity.
Time Frame: at autopsy within 9 months of baseline scan
Population: Autopsy cohort N=64. n=39 were truth positive for NFTs. n=25 were truth negative for NFTs.
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Sensitivity of Flortaucipir vs Autopsy NFT Score B3: Subjects with a truth positive NFT Score (B3)
- Specificity of Flortaucipir vs Autopsy NFT Score <B3: Subjects with a truth negative NFT Score (B2 or lower)
Arm/Group | Sensitivity of Flortaucipir vs Autopsy NFT Score B3 | Specificity of Flortaucipir vs Autopsy NFT Score <B3
Number analyzed (Participants) | 39 | 25
percentage of cases correctly identified | 92.3 [79.7 to 97.3] | 80.0 [60.9 to 91.1]

4. Secondary Outcome: Flortaucipir Diagnostic Performance (NIA-AA Autopsy Diagnosis)
Description: Sensitivity and specificity of majority interpretation of of AD pattern tau PET scan corresponding to NIA-AA autopsy diagnosis. The 95% CIs provided for specificity and sensitivity were based on the Wilson score method. The hypothesis tested was that majority read results had the lower bound of the 2-sided 95% CI greater than or equal to 55% for both sensitivity and specificity.
Time Frame: at autopsy within 9 months of baseline scan
Population: Autopsy cohort N=64. n=38 were truth positive for NFTs. n=26 were truth negative for NFTs.
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Sensitivity Majority Read NIA-AA Autopsy Diagnosis: Subjects with a truth positive NIA-AA autopsy diagnosis (High ADNC)
- Specificity Majority Read NIA-AA Autopsy Diagnosis: Subjects with truth negative NIA-AA autopsy diagnosis (No/Low/Intermediate ADNC)
Arm/Group | Sensitivity Majority Read NIA-AA Autopsy Diagnosis | Specificity Majority Read NIA-AA Autopsy Diagnosis
Number analyzed (Participants) | 38 | 26
percentage of cases correctly identified | 94.7 [82.7 to 98.5] | 80.8 [62.1 to 91.5]

5. Secondary Outcome: Inter-Reader Agreement
Description: Fleiss' Kappa statistics were used to assess inter-reader agreement for the diagnostic decisions associated with primary outcome 1. Fleiss' kappa is a statistical measure for assessing the reliability of agreement between a fixed number of raters when assigning categorical ratings to a number of items or classifying items. Fleiss' kappa can range from 0 to 1 with 1 indicating perfect agreement between the readers. Results are reported as overall agreement, calculated as proportion of scans where reader pairs agreed, divided by the total number of scans read by each reader pair.
Time Frame: baseline scan
Measure: Number; unit: proportion of agreed cases
Groups:
- All Cases Read: All participants from the study for which a visual read flortaucipir PET result was obtained (n=105), regardless of whether the subject had a valid autopsy
Arm/Group | All Cases Read
Number analyzed (Participants) | 105
proportion of agreed cases
  Reader 1 v Reader 2 | 0.79
  Reader 1 v Reader 3 | 0.79
  Reader 1 v Reader 4 | 0.79
  Reader 1 v Reader 5 | 0.81
  Reader 2 v Reader 3 | 0.96
  Reader 2 v Reader 4 | 0.88
  Reader 2 v Reader 5 | 0.65
  Reader 3 v Reader 4 | 0.92
  Reader 3 v Reader 5 | 0.68
  Reader 4 v Reader 5 | 0.72
Statistical Analysis 1: Comparison: All Cases Read; Inter-reader agreement analysis using Fleiss' kappa. The hypothesis tested was that the observed kappa values were ≥0.64 and the lower bound of the 2-sided 95% CIs were ≥0.55 for the inter-reader agreement among readers; Test type: Other; Fleiss' kappa = 0.80, 95% CI 2-sided [0.74 to 0.86]

6. Other Pre Specified Outcome: Diagnostic Performance of Individual Readers (NFT Score B2-B3 as Truth Positive)
Description: Sensitivity and specificity of 5 independent readers' interpretations of ante-mortem flortaucipir PET imaging for detection of a pattern of flortaucipir neocortical uptake that corresponds to neurofibrillary tangles (NFT) Score of B3 (Hyman et al., 2012; Montine et al., 2012). NFT B scores range from B0 (no NFTs in the brain) to B3 (widespread NFTs in the brain). Sensitivity and specificity are percentages that can range from 0 to 100%. For this analysis, B scores of B2-B3 were considered truth positive, and B scores of B0-B1 were considered truth negative.
Time Frame: at autopsy within 9 months of baseline scan
Population: Autopsy cohort N=64. n=56 were truth positive for NFTs. n=8 were truth negative for NFTs.
Measure: Number (95% Confidence Interval); unit: percentage of cases correctly identified
Groups:
- Sensitivity of Flortaucipir vs Autopsy NFT Score B2-B3: Subjects with a positive autopsy NFT score truth standard (NFT B2 or B3)
- Specificity of Flortaucipir vs Autopsy NFT Score B0-B1: Subjects with a negative autopsy NFT score truth standard (NFT B0 or B1)
Arm/Group | Sensitivity of Flortaucipir vs Autopsy NFT Score B2-B3 | Specificity of Flortaucipir vs Autopsy NFT Score B0-B1
Number analyzed (Participants) | 56 | 8
percentage of cases correctly identified
  Reader 1 | 80.4 [68.2 to 88.7] | 87.5 [52.9 to 97.8]
  Reader 2 | 67.9 [54.8 to 78.6] | 100.0 [67.6 to 100.0]
  Reader 3 | 67.9 [54.8 to 78.6] | 87.5 [52.9 to 97.8]
  Reader 4 | 73.2 [60.4 to 83.0] | 87.5 [52.9 to 97.8]
  Reader 5 | 85.7 [74.3 to 92.6] | 62.5 [30.6 to 86.3]

ADVERSE EVENTS:
Time Frame: 9 months after flortaucipir scan, up to a total of 18 months if a subject was re-scanned per protocol
Description: Adverse events (AEs) were collected at scan visits, regardless of attribution to study drug. End of study for AE reporting was 48 hours after the last study drug administration. AEs occurring after study drug administration, but outside that window were not recorded, unless considered attributable to study drug.
Groups:
- Safety Analysis Population: All enrolled subjects from the flortaucipir PET scan arm who received one dose of flortaucipir
Arm/Group | Safety Analysis Population
All-Cause Mortality (participants affected / at risk) | 73/156
Serious Adverse Events (participants affected / at risk) | 3/156
Other Adverse Events (participants affected / at risk) | 14/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Population (N=156)
acute kidney injury (Renal and urinary disorders) | 1 (1)
malignant neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
myocardial infarction (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Analysis Population (N=156)
myocardial infarction (Cardiac disorders) | 1 (1)
vertigo (Ear and labyrinth disorders) | 1 (1)
diarrhoea (Gastrointestinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 1 (1)
injection site bruising (General disorders) | 1 (1)
fall (Injury, poisoning and procedural complications) | 1 (1)
procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1)
myopathy (Musculoskeletal and connective tissue disorders) | 1 (1)
headache (Nervous system disorders) | 2 (2)
dizziness postural (Nervous system disorders) | 1 (1)
hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
tremor (Nervous system disorders) | 1 (1)
agitation (Psychiatric disorders) | 3 (3)
mental disorder (Psychiatric disorders) | 1 (1)
restlessness (Psychiatric disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2017-12-18): https://cdn.clinicaltrials.gov/large-docs/46/NCT02516046/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT02516046/SAP_001.pdf